CLINICAL TRIAL: NCT04805437
Title: 3D Designed Boston Brace Versus Standard Boston Brace in Halting Progression in Idiopathic Scoliosis: a Randomized Controlled Trial
Brief Title: Brace Treatment for Idiopathic Scoliosis; PReventing Idiopathic SCOliosis PROgression
Acronym: PRISCOPRO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Paul Gerdhem, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ED-PG-AA-2021-Brace
Record Dates: First submitted 2021-03-13; First posted 2021-03-18 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Idiopathic Scoliosis
Keywords: Idiopathic scoliosis; Randomized controlled trial; Brace; Orthosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Orthotist and research nurse will know what type of brace the participant receives, but will not tell the participant which type he/she has received. Investigators, care providers and outcome assessors will be blinded for type of brace.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D TLSO (Experimental): A 3-dimensional Boston brace will be designed to the patient's individual type of scoliosis. In-brace radiographs will be performed after prescription. Reinforcement of the assigned intervention will be performed in conjunction with reassessment every 6 months. Patients are encouraged to use the brace for 20 hours per day and to also continue with physical activities for the entirety of the study. Compliance will be monitored with a heat sensor built in the brace that measures wearing time.
  Interventions: Device: 3D TLSO
- Standard TLSO (Active Comparator): A standard Boston brace will be designed to the patient's individual type of scoliosis. In brace radiographs will be performed after prescription. Reinforcement of the assigned intervention will be performed in conjunction with reassessment every 6 months. Patients are encouraged to use the brace for 20 hours per day and to also continue with physical activities for the entirety of the study. Compliance will be monitored with a heat sensor built in the brace that measures wearing time.
  Interventions: Device: Standard TLSO

INTERVENTIONS:
Device: 3D TLSO — Brace treatment with Boston 3D 20 hours a day until skeletal maturity.
  Other Names: Boston 3D brace
  Arms: 3D TLSO
Device: Standard TLSO — Brace treatment with standard Boston brace 20 hours a day until skeletal maturity.
  Other Names: Boston brace
  Arms: Standard TLSO

SUMMARY:
Idiopathic scoliosis is the most common spinal deformity in children and adolescents with an estimated prevalence of 3%. About one tenth of the children with scoliosis develop a deformity that requires treatment with brace or surgery with the current treatment protocol. When brace treatment for scoliosis is indicated, standard treatment consists of bracing 20 hours or more per day. Outcomes of brace treatment depend to a large extent on wearing time and since many adolescents feel uncomfortable in the brace, it is of importance to combine efficacy and comfortability of the brace.

DETAILED DESCRIPTION:
Bracing with a rigid TLSO is gold-standard treatment in terms of halting progression of idiopathic scoliosis in skeletally immature adolescents and children. The treatment is cumbersome and demanding for adolescents during a vulnerable stage in life, and may be associated with poor compliance. Furthermore, the treatment lasts in many cases for several years and has shown to have a negative psychological effect for patients. Since time in brace is of utmost importance for best possible outcome, the braces need to be tolerated by the patients. As of today, 3D designed braces have received much attention and are thought to increase comfortability and ultimately increase wearing time, leading to better outcomes.

In a multicenter randomized controlled trial, we seek to compare standard Boston brace to a newly developed 3D designed Boston brace. Skeletally immature patients with idiopathic scoliosis will be randomized to receive either standard Boston brace or Boston 3D brace. All patients will be encouraged to be physically active for 60 minutes per day. Patients, outcome assessors and clinician in charge during follow-ups will be blinded for the type of brace the patients are being treated with. Thermal sensors will be installed in all braces to monitor compliance. Outcome include change in curve severity, quality of life and surgical rates. Patients will be evaluated with clinical and radiological follow-ups every six months until skeletal maturity and thereafter at 2, 5 and 10 years. Curve progression will not lead to change of brace. A total of 85 individuals are required in each group based on the hypothesis of a 2% failure rate in the 3D-brace group and 15% in the standard brace group with 5% significance level and 80% power and consideration for dropout of up to 20%.

For individuals who are not willing to be randomized and participate in the study, standard Boston brace will be offered and these individuals will serve as an observational group with similar follow-ups and will be asked to answer same survey as the study populations will do.

ELIGIBILITY:
Inclusion Criteria:

* Cobb 25-40 degrees
* Skeletally immature, Sanders score of 6 or less and Risser 2 or less.
* Menarche status maximum one year in females
* Aged 9-17 years
* No previous brace treatment or surgery for scoliosis
* Apex of the primary curve at T7 or caudal

Exclusion Criteria:

* Non-idiopathic scoliosis (i.e. neuromuscular, syndromic or congenital scoliosis)
* Previous spine surgery

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 170 (Estimated)
Dates: Start 2021-04-30 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2037-04 (Estimated)

PRIMARY OUTCOMES:
Curve progression | Measured at each six-month follow-up until skeletal maturity. Skeletal maturity defined as less than 1 cm body height increase in 6 months.
  Increase in curve severity (Cobb angle) of more than 6 degrees on two consecutive radiographs after baseline

SECONDARY OUTCOMES:
Clinical outcomes | At each six-month follow-up and 2, 5, 10 years after skeletal maturity
  Angle of trunk rotation in forward bending, assessed with scoliometer
Patient-reported outcome measures | At each six-months follow-up and 2, 5, 10 years after skeletal maturity
  Scoliosis Research Society-22r questionnaire
Patient-reported outcome measures | At each six-month follow-up, and 2, 5, 10 years after skeletal maturity
  EQ5D questionnaire
Patient-reported outcome measures | At each six-month follow-up, and 2, 5, 10 years after skeletal maturity
  Spinal Appearance Questionnaire (SAQ)
Patient-reported outcome measures | At each six-month follow-up, and 2, 5, 10 years after skeletal maturity
  International Physical Activity Questionnaire (IPAQ)
Surgical rates | At each six-months follow-up and 2, 5, 10 years after skeletal maturity
  Number needing surgical intervention

CONTACTS AND LOCATIONS:
Overall Officials: Elias Diarbakerli, PT, PhD, Principal Investigator — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Linköping university hospital, Linköping
  - Karolinska university hospital, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
IPD underlying published manuscripts will be accessible for other researchers.
Supporting Information: Study Protocol, SAP
Time Frame: The study protocol will be submitted to a peer-reviewed journal.
Access Criteria: The investigators in charge will be responsible for reviewing access requests. Crude data, randomization procedures and intervention details can be shared with other researchers upon request.

REFERENCES:
- [Derived] Diarbakerli E, Charalampidis A, Abbott A, Gerdhem P. PReventing Idiopathic SCOliosis PROgression (PRISCOPRO): A protocol for a quadruple-blinded, randomized controlled trial comparing 3D designed Boston brace to standard Boston brace. PLoS One. 2021 Aug 9;16(8):e0255264. doi: 10.1371/journal.pone.0255264. eCollection 2021. PMID 34370760